CLINICAL TRIAL: NCT03230903
Title: Physical Telerehabilitation in Patients With Multiple Sclerosis With Significant Mobility Impairment
Brief Title: Physical Telerehabilitation in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joel Stein, MD, Simon Baruch Professor of Physical Medicine & Rehabilitation, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAQ7693; MS150167 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-01-04; First posted 2017-07-27 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Telerehabilitation; Physical rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home Telerehabilitation (Experimental): The physical telerehabilitation group will receive an exercise plan, exercise equipment, a computer, and access to a daily individualized exercise plan. Participants in this group will follow the exercise plan that is sent to their computer via the telerehabilitation software. Participants will have interactions with a physical therapist and an exercise physiologist throughout training intervention.
  Interventions: Other: Home telerehabilitation
- Usual Care (Sham Comparator): The usual care group will receive an individualized exercise program at baseline however participants will not receive the home telerehabilitation system or exercise equipment. Participants assigned to the usual care group will also not have access to the study physical therapist or exercise physiologist during the intervention.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Home telerehabilitation — Patients will receive an individualized exercise plan sent to a computer at their home. Patients will have daily access to a physical therapist and exercise physiologist.
  Arms: Home Telerehabilitation
Other: Usual Care — Patients will receive a written individualized exercise plan during their baseline visit on top of their usual disease care.
  Arms: Usual Care

SUMMARY:
The study aims to evaluate the efficacy of the MS HAT (Multiple Sclerosis Home Automated Telemanagement) System as an adjunct to the current standard of medical care for patients with MS (PwMS). The individual patient with MS will be the unit of analysis. For each participant, the investigators will assess the effect of Home Automated Telemanagement (HAT) on functional outcomes, levels of disablement including impairment, activity and participation, socio-behavioral parameters, and satisfaction with medical care as described below.

DETAILED DESCRIPTION:
People with multiple sclerosis may develop severe disability over the time. Physical therapy including regular exercise helps patients with severe disability to maintain muscle strength, reduce disease symptoms and improve quality of life. However physical therapy programs at clinical settings require constant travel which may limit access of patients with mobility disability to these services on continuous basis.Technology can allow patients with mobility disability exercise at home under supervision of their rehabilitation team. Currently it is unclear how effective this approach is. The study aims to demonstrate that the patients who were helped by the new technology to exercise at home will have better fitness, less symptoms and better quality of life. If so, other patients with significant mobility disability will be able to take advantage of this technology. This approach can be extended to people with different diseases causing mobility impairment and it can be used not only for physical but also for cognitive and occupational rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age >21
* Confirmed diagnosis of Multiple Sclerosis based on McDonald criteria
* EDSS range 5.0-8.0
* Mini-Mental State Examination (MMSE) > 22 or presence of a caregiver to assist in daily exercise regimen

Exclusion Criteria:

* Coronary artery disease
* Congestive Heart Failure
* Uncontrolled hypertension
* Epilepsy
* Pacemaker or implanted defibrillator
* Unstable fractures or other musculoskeletal diagnoses

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-10; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Baseline up to 6 months
  Cardiorespiratory fitness will be measured by oxygen consumption

SECONDARY OUTCOMES:
MS Self-efficacy scale | Baseline up to 6 months
  MS Self-efficacy scale is a 14-point questionnaire designed to assess the psychological adjustment and quality-of-life of individuals with MS.
Exercise adherence | Baseline up to 6 months
  Exercise adherence will be measured by the number of sessions completed by the participant out of the number of exercise sessions prescribed.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline up to 6 months
  The CES-D is a 20 point questionnaire based on self-reported frequency of symptoms related to depression during the past week.
Berg Balance Scale (BBS) | Baseline up to 6 months
  BBS is a clinical 14-item scale designed to measure balance
2-Minute Walk Test (2MWT) | Baseline up to 6 months
  Total distance walked in meters will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided